CLINICAL TRIAL: NCT02095743
Title: Phase II Randomised Study Comparing the Tolerance of PICC Line (Peripherally Inserted Central Catheter) and Implanted Port for Adjuvant Chemotherapy in HER2-negative Early Breast Cancer
Brief Title: Tolerance of PICC Line Versus Implanted Port for Adjuvant Chemotherapy in Early Breast Cancer
Acronym: EPIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHB 13-01
Record Dates: First submitted 2013-10-25; First posted 2014-03-26 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Early Stage Breast Carcinoma
Keywords: Early breast cancer; Chemotherapy; PICC line; Implanted port
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PICC line (Experimental): Use of a PICC line for chemo administration (PowerPICC SOLO²)
  Interventions: Device: Use of a PICC line for chemo administration (PowerPICC SOLO²)
- Implanted Port (Active Comparator): Use of an implanted port for chemo administration
  Interventions: Device: implanted port for chemo administration (X-port isp); Device: Use of a PICC line for chemo administration (PowerPICC SOLO²)

INTERVENTIONS:
Device: implanted port for chemo administration (X-port isp)
  Other Names: X-port isp M.R.I Implantable Port (Bard Access Systems Inc)
  Arms: Implanted Port
Device: Use of a PICC line for chemo administration (PowerPICC SOLO²) — The description of the device could found on the published marketing authorisation
  Other Names: kit PowerPICC SOLO² (Bard Access Systems Inc)

SUMMARY:
Adjuvant chemotherapy is frequently proposed to patients presenting early breast cancer, in case of high risk of recurrence (large tumors, node involvement, high grade…). Due to its toxicity toward veins, chemotherapy must be administered through a central venous device. Today, one can use either an implanted port or a PICC line (Peripherally Inserted Central Catheter). A PICC line is easier to implant and to explant, but has to be flushed every week and may impact daily life (no swimming, some clothes may not fit). On the other hand, a port is subcutaneous and lets patients lead a normal life, but its implant and explant require a cutaneous incision with possible complications (bleeding, pain, infection). For both venous devices, complications such as thrombosis or infection may happen. Published data comparing the two devices are heterogeneous and do not often distinguish patients treated for different diseases at various stages. Empirically in daily practice, for long term use (>6 months) a port is usually preferred, whereas for short-term treatments (<6 weeks) a PICC line is used. In the case of Her2 negative early breast cancer, adjuvant chemotherapy usually lasts 4 to 5 months. There is no scientific evidence for preferring one device to the other for these patients.

The aim of this study is to prospectively compare the patients' satisfaction and tolerance of each of the two devices.

DETAILED DESCRIPTION:
The intravenous device will be randomly attributed. The adjuvant chemotherapy regimen will be selected according the standards of the center ( 6 cycles of FEC100 or 3 cycles of FEC100 then 3 cycles of Taxotere (docetaxel). The patient will be followed as per center's standards and visits (prior, during and after every drug administration, then monthly for six months). All Adverse Events will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Women age > 18
* Documented breast cancer
* No Her2 overexpression
* Patients operated with curative intent (no distant metastasis at diagnosis)
* Patients undergoing an adjuvant chemotherapy consisting of 3 courses of FEC 100 (5-fluorouracil, epirubicin 100mg/m² and cyclophosphamide ) followed by 3 courses of Taxotere, or 6FEC100 (according to CHB refencial for localised breast cancer treatment).
* Signed informed consent

Exclusion Criteria:

* Bilateral axillary node dissection
* History of bilateral upper thoracic irradiation
* Cutaneous disease (eczema, scleroderma, infection…) at catheter insertion site (arm or upper thorax)
* Recent thrombosis of the upper body
* Therapeutic anticoagulation
* Tracheotomy
* Treatment for bacteriemia in process
* Altered hemostasis: INR > 1.5 ; APTT > 1.5 , platelets < 60 G/l
* Renal failure with creatinine clearance < 60mL/min
* Involvement in another trial
* Contraindication to chemotherapy by FEC 100 or taxotere
* Pregnancy or breast feeding
* Protected major patient (under guardianship).
* Psychosocial disorders : decompensated mental disorders, no social security coverage, patient who does not speak french

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Probability of occurrence of a significant adverse event related to the central venous device | 37 weeks
  To define between the two device (PICC line and implanted port) which one provides the less probability of occurrence of a significant adverse event related to the device (SAERD), from the insertion to the first consultation of survey (36-38 weeks after implantation of the device which is also 5 months after its ablation).

SECONDARY OUTCOMES:
Patients' satisfaction for the use of their central venous device | 1 year
  Evaluation of the patients' satisfaction assessed by the QLQ C30, and by a 19 questions home-made questionnaire dedicated to the use of central veinous devices

CONTACTS AND LOCATIONS:
Overall Officials: Florian Clatot, MD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

REFERENCES:
- [Derived] Lefebvre L, Noyon E, Georgescu D, Proust V, Alexandru C, Leheurteur M, Thery JC, Savary L, Rigal O, Di Fiore F, Veyret C, Clatot F. Port catheter versus peripherally inserted central catheter for postoperative chemotherapy in early breast cancer: a retrospective analysis of 448 patients. Support Care Cancer. 2016 Mar;24(3):1397-403. doi: 10.1007/s00520-015-2901-8. Epub 2015 Sep 5. PMID 26342484